CLINICAL TRIAL: NCT00361270
Title: Treatment of Veterans With Chronic Low Back Pain
Acronym: CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D4421-I; H-18610 (Other: Baylor College of Medicine IRB)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Results first posted 2015-08-26 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Low Back Pain, Recurrent
Keywords: Biofeedback; Hypnosis; Low Back Pain, Recurrent; Pain beliefs; Pain coping strategies; Pain intensity; Pain interference; Pain quality; Self-help treatment; Sleep dysfunction
MeSH Terms: conditions — Low Back Pain; Pain; Parasomnias | interventions — bradykinin, Hyp(3)-TyrMe(8)-; DMAC2L protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 Hyp-8 (Experimental): Single-site study at MEDVA-Houston Behavioral: 8 weeks 1-hour hypnosis with hypnotherapist without audio recordings
  Interventions: Behavioral: Hyp-8
- Arm 2 Hyp-8 w recordings (Experimental): Single-site study at MEDVA-Houston Behavioral: 8 weeks 1-hour hypnosis with hypnotherapist with audio recordings
  Interventions: Behavioral: Hyp-2 w recordings; Behavioral: Hyp-8; Behavioral: Hyp-8 w recordings
- Arm 3 Hyp-2 w recordings (Experimental): Single-site study at MEDVA-Houston Behavioral: 2 weeks 1-hour hypnosis with hypnotherapist with audio recordings
  Interventions: Behavioral: Hyp-2 w recordings; Behavioral: Hyp-8; Behavioral: Hyp-8 w recordings
- Arm 4 BIO (Active Comparator): Single-site study at MEDVA-Houston Behavioral: 8 weeks 1-hour EMG biofeedback without audio recordings
  Interventions: Behavioral: BIO

INTERVENTIONS:
Behavioral: Hyp-8 — 8 weekly 1-hour sessions of therapist-guided hypnosis
  Other Names: Arm 1
  Arms: Arm 1 Hyp-8
Behavioral: Hyp-2 w recordings — 2 weeks of 1-hour sessions of therapist-guided hypnosis + 6 weeks of daily home practice with hypnosis CDs
  Other Names: Arm 3
  Arms: Arm 2 Hyp-8 w recordings
Behavioral: Hyp-8 — 8 weekly 1-hour sessions of therapist-guided hypnosis
  Other Names: Arm 1
  Arms: Arm 2 Hyp-8 w recordings
Behavioral: Hyp-8 w recordings — 8 weekly 1-hour sessions of therapist-guided hypnosis + daily home practice with hypnosis CDs
  Other Names: Arm 2
  Arms: Arm 2 Hyp-8 w recordings
Behavioral: Hyp-2 w recordings — 2 weeks of 1-hour sessions of therapist-guided hypnosis + 6 weeks of daily home practice with hypnosis CDs
  Other Names: Arm 3
  Arms: Arm 3 Hyp-2 w recordings
Behavioral: Hyp-8 — 8 weekly 1-hour sessions of therapist-guided hypnosis
  Other Names: Arm 1
  Arms: Arm 3 Hyp-2 w recordings
Behavioral: Hyp-8 w recordings — 8 weekly 1-hour sessions of therapist-guided hypnosis + daily home practice with hypnosis CDs
  Other Names: Arm 2
  Arms: Arm 3 Hyp-2 w recordings
Behavioral: BIO — 8 weekly 1-hour sessions of EMG Biofeedback without hypnotic suggestion
  Other Names: Arm 4
  Arms: Arm 4 BIO

SUMMARY:
The purpose of this study is to assess the effectiveness of hypnosis in the treatment of chronic low back pain.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is one of the most disabling and common conditions (Loeser, 2001). Eighty percent of men and women will suffer from acute back pain at some point in their lives, with an estimated 10% becoming chronic (King et al., 2001); and the cost of CLBP to society is staggering (Turk, 2002). For example, a nation-wide study of the VHA Health Care System by Yu and colleagues (Yu et al., 2003) reported that 10.6% or 361,868 Veterans who were being cared for by the VA suffered from CLBP, costing the system an estimated $22 million dollars in fiscal year 1999 alone. This figure applies to the cost of medical care only and does not include the cost from the impact of the condition on the Veterans such as disability, lost wages, and other associated medical and psychiatric conditions as well as untold suffering and interference in daily activities.

The efficacy of hypnosis as a treatment for acute and some chronic pain conditions has been well documented. One recent meta-analysis of 18 studies indicated a moderate to large hypno-analgesic effect (Montgomery et. al., 2000). Included in this meta-analysis were studies of a variety of clinical pain syndromes, such as acute/transient pain resulting from burns, radiological procedures, or coronary/ischemic pain, as well as chronic pain due to cancer or headaches. However, none of the studies in this review targeted CLBP. The authors concluded that ".the average participant treated with hypnosis demonstrated greater analgesic response than 75% of participants in standard and no-treatment groups" (page 143). Similarly, Patterson and Jensen (2003) reviewed randomized control trials of hypnosis and clinical pain, and concluded that "Hypnosis has a reliable and significant impact on acute procedural pain and chronic pain conditions."

The proposed research will (1) conduct a randomized controlled clinical trial to further validate and confirm the findings from a recently completed pilot project showing that hypnosis is efficacious in reducing pain intensity and pain interference and the improving the quality of life of Veterans suffering from CLBP (see preliminary studies section, below), (2) evaluate the relative importance of home practice of hypnosis, (3) determine if the beneficial effects of hypnosis are long lasting, and (4) determine the predictors of treatment outcome, in particular, hypnotizability (a general and stable trait ability to respond to hypnotic suggestions), but also frequency of practice. In this study, a control condition will be used that is credible to patients, but is known to have only minimal effects on pain.

The four treatment groups are: Group 1 - full in-person hypnosis series (8 sessions) without home practice, Group 2 - full in-person hypnosis series (8 sessions) with home practice with CDs, Group 3 - brief in-person hypnosis series (2 sessions) with home practice with CDs, and Group 4 - a minimally effective control condition (minimal biofeedback (8 sessions) designed to appear credible but have minimal effects). Subjects: 160 subjects will be recruited from the MEDVAMC Pain Management Program via posters and the program staff. Inclusion criteria: Chronic low back pain for at least 6 months, pain severity at least 5 on a 0-10 scale, and pain is primarily musculoskeletal/mechanical. Exclusion criteria: Acute and cancer pain, neuropathic etiology, severe psychopathology, active substance abuse, significant cognitive deficit, and previous participant of the pilot study on hypnosis and chronic low back pain. Outcome measures that will be administered pre- and post-intervention include: Brief Pain Inventory, Numeric Rating Scale, Pittsburgh Sleep Quality Scale, McGill Pain Questionnaire, Pain Quality Assessment Scale, Rand MHI-5, Hypnosis Treatment Outcome Measure, and the Two-Item Measures of Pain Beliefs and Coping Strategies. A process measure is the frequency of home practice.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain for at least 6 months
* Pain severity at least 5 on a 0-10 scale
* Pain is primarily musculoskeletal/mechanical
* Adults, at least 18 years of age

Exclusion Criteria:

* Acute and cancer pain
* Neuropathic etiology
* Severe psychopathology
* Active substance abuse
* Significant cognitive deficit
* Previous participant of the pilot study on hypnosis chronic low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2010-02-15 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wright Williams, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypnosis-8: 8 sessions of hypnosis with no practice cds
- Hypnosis-Practice 8: 8 sessions hypnosis with practice cds
- Hypnosis Practice 2: 2 sessions of hypnosis with practice cds
- Biofeedback - 8: 8 sessions biofeedback
Period: Overall Study
Arm/Group | Hypnosis-8 | Hypnosis-Practice 8 | Hypnosis Practice 2 | Biofeedback - 8
Started | 49 | 39 | 35 | 38
Completed | 25 | 25 | 25 | 25
Not Completed | 24 | 14 | 10 | 13
Not completed — Death | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 4 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 9 | 4 | 5 | 4
Not completed — Withdrawal by Subject | 6 | 6 | 3 | 7
Not completed — Afraid of Hypnosis | 1 | 2 | 0 | 0
Not completed — Problems with Transportation | 4 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Single-site study at MEDVA-Houston
  Therapist-guided hypnosis: 8 weekly 1-hour sessions of therapist-guided hypnosis
- Arm 2: Single-site study at MEDVA-Houston
  Therapist-guided hypnosis: 8 weekly 1-hour sessions of therapist-guided hypnosis with home practice with hypnosis CDs
- Arm 3: Single-site study at MEDVA-Houston
  Home practice with hypnosis CDs: 2 weeks of 1-hour sessions of therapist-guided hypnosis + 6 weeks of daily home practice with hypnosis CDs
- Arm 4: Single-site study at MEDVA-Houston
  EMG Biofeedback without hypnotic suggestion: 8 weekly 1-hour sessions of EMG Biofeedback without hypnotic suggestion
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 49 | 39 | 35 | 38 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 33 | 30 | 33 | 136
  >=65 years | 9 | 6 | 5 | 5 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 8 | 8 | 31
  Male | 42 | 31 | 27 | 30 | 130
BPI Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — This is a 4 item scale. Each item measures pain on a 0-10 No pain - Worst pain scale. The overall measure ranges from 0 to 40.
  units on a scale | 24.28 (5.44) | 24.50 (5.52) | 21.08 (5.14) | 25.50 (6.05) | 24.37 (6.26)
BPI Interference [Mean (Standard Deviation); unit: units on a scale] — This is a 10 item scale. Each item measures pain on a 0-10 No pain - Worst pain. The overall scale values range from 0 to 100.
  units on a scale | 61.20 (17.55) | 52.06 (19.62) | 49.60 (20.65) | 11.36 (3.55) | 56.15 (20.15)
PSQI [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) contains19 items with 7 component scores ranging from 0 no difficulty falling asleep to 3 severe difficulty. Component scores are then added to create a global score ranging from 0 no difficulty falling asleep to 21 severe difficulty falling asleep.
  units on a scale | 11.36 (3.55) | 11.80 (4.08) | 9.68 (4.15) | 10.24 (4.02) | 11.16 (4.17)

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-Treatment to 1-week Post Treatment on Brief Pain Inventory-Pain Intensity Scale
Description: The change score measures the difference between Pre-Treatment Brief Pain Inventory Pain Intensity Scale scores (Numerical Rating Scale (NRS): 0 no pain - 10 worst pain) and the 1-week Post--Treatment Brief Pain Inventory-Pain Intensity Scale scores for 4 items. Change is calculated as pre-treatment minus post treatment.
Time Frame: Subjects change on this scale from Pre-Treatment to 1 week post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hypnosis-8: 8 1-hour sessions of hypnosis without audio recordings
- Hypnosis-Practice 8: 8 1-hour sessions of hypnosis with audio recordings
- Hypnosis Practice 2: 2 1-hour sessions of hypnosis with audio recordings
- Biofeedback - 8: 8 1-hour sessions of EMG biofeedback
Arm/Group | Hypnosis-8 | Hypnosis-Practice 8 | Hypnosis Practice 2 | Biofeedback - 8
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale | 17.52 (10.24) | 14.16 (8.78) | 13.78 (9.04) | 21.18 (9.22)

2. Secondary Outcome: Change From Pre-treatment to 1- Week Post Treatment on Brief Pain Inventory-Interference Scale
Description: The change score measures the difference between pre-treatment scores on the Brief Pain Inventory-Interference Scale (NRS: 0 no interference - 10 complete interference) and 1- week post treatment scores for the 10 items. Change is calculated as pre-treatment minus post treatment.
Time Frame: Subjects change on this scale from Pre-Treatment to 1-week post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hypnosis-8: 8 1-hour sessions of hypnosis with hypnotherapist without recordings
- Hypnosis-Practice 8: 8 1-hour sessions with hypnotherapists with audio recordings
- Hypnosis Practice 2: 2 1-hour sessions with hypnotherapist with audio recordings
- Biofeedback - 8: 8 1-hour sessions of EMG biofeedback without recordings
Arm/Group | Hypnosis-8 | Hypnosis-Practice 8 | Hypnosis Practice 2 | Biofeedback - 8
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale | 39.08 (29.39) | 31.88 (25.66) | 29.00 (25.99) | 45.4 (23.67)

3. Secondary Outcome: Change From Pre Treatment to 1-week Post Treatment on Pittsburgh Sleep Quality Index (PSQI)
Description: The change score is the difference between pre-treatment scores on the Pittsburgh Sleep Quality Index (PSQI) and the 1-week post-treatment scores. Positive values indicate a reduction in sleep problems. The PSQI was scored on 19 items with 7 component scores ranging from 0 no difficulty falling asleep to 3 severe difficulty, then component scores added to create global score ranging from 0 no difficulty falling asleep to 21 severe difficulty falling asleep.
Time Frame: Subjects change on this scale from Pre-treatment to 1-week post treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hypnosis-Practice 8: 8 1-hour sessions with hypnotherapist and audio recordings
- Hypnosis Practice 2: 2 1-hour sessions with hypnotherapist and audio recordings
- Biofeedback - 8: 8 1-hour sessions of EMG biofeedback no recordings
Arm/Group | Hypnosis-8 | Hypnosis-Practice 8 | Hypnosis Practice 2 | Biofeedback - 8
Number analyzed (Participants) | 25 | 25 | 25 | 25
units on a scale | 9.96 (4.37) | 8.72 (4.31) | 7.8 (4.92) | 8.88 (3.99)

ADVERSE EVENTS:
Groups:
- Hypnosis-8: 8 1-hour sessions with hypnotherapist
- Hypnosis-Practice 8: 8 1-hour sessions with hypnotherapist with audio recordings
Arm/Group | Hypnosis-8 | Hypnosis-Practice 8 | Hypnosis Practice 2 | Biofeedback - 8
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/39 | 0/35 | 0/38
Other Adverse Events (participants affected / at risk) | 0/49 | 1/39 | 1/35 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypnosis-8 (N=49) | Hypnosis-Practice 8 (N=39) | Hypnosis Practice 2 (N=35) | Biofeedback - 8 (N=38)
Nightmares (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Nightmares
Disturbing Images (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Disturbing images and thoughts

LIMITATIONS AND CAVEATS:
The study is done on a population of Veterans and may not generalize to the larger population. The same provider administered treatment for all four groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes